CLINICAL TRIAL: NCT07267715
Title: EVA: Evaluation of EVOKE Therapy Metrics Generated Using the Evoke System With EVA
Status: Not yet recruiting | Type: Observational
Sponsor: Dustin Reynolds, MD (Other)
Collaborators: Saluda Medical Pty Ltd (Industry)
Responsible Party: Sponsor-Investigator, Dustin Reynolds, MD, Interventional Pain Management Specialist, Anesthesiologist, Mount Carmel Health System
Organization: Mount Carmel Health System (Other)
Other Study IDs: 250714-1
Record Dates: First submitted 2025-11-18; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Chronic Pain
Keywords: Treatment of chronic pain of the trunk and/or limbs.
MeSH Terms: conditions — Chronic Pain | interventions — Spinal Cord Stimulation; Drug Delivery Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- SCS Evoke System Implant: Subjects with chronic, intractable focal pain of the trunk and/or limbs who undergo Evoke System implant.
  Interventions: Device: Spinal Cord Stimulation (SCS) System

INTERVENTIONS:
Device: Spinal Cord Stimulation (SCS) System — Spinal cord stimulation system as an aid in the management of chronic intractable pain of the trunk and/or limbs; and will be used within its commercially approved indication.

SUMMARY:
The Evoke Spinal Cord Stimulator (SCS) System (Evoke® System) is an FDA-approved device that is used to manage long lasting, severe pain that is not relieved by typical medical treatments.

This research registry is being conducted to collect data from patients treated with a SCS device in order to determine how the device impacts their chronic pain condition.

Specifically, the study aims to:

* Evaluate data collected from the SCS system on how well the system is working.
* Evaluate the feasibility of programming the SCS system independently without external assistance.
* Evaluate changes in physical function, fatigue, pain interference, mood, sleep, daily activities, pain control, and overall satisfaction with the device.

ELIGIBILITY:
Inclusion Criteria:

* Subject is not pregnant and 18 years of age or older at the time of enrollment.
* Subject has a minimum NRS score of 6 or higher (where 10 indicates the worst imaginable pain) in primary area of pain at baseline.
* Subject is planning to have a temporary trial with the Evoke® System to aid in the management of chronic intractable pain of the trunk and/or limbs.
* Subject is willing to program the Evoke® System using EVA™ under the supervision of the study investigator or Qualified Health Professional.
* Subject is being trialed with a neurostimulation system for the first time.
* Subject is able to read and understand English.
* Subject is capable of subjective evaluation; subject must be able to describe and rate his/her pain levels.
* Subject is willing and capable of giving informed consent.
* Subject is willing and able to comply with study-related requirements, procedures, and visits.
* Subject has adequate cognitive ability to use a patient programmer and recharger as determined by the Investigator.

Exclusion Criteria:

- There are no exclusion criteria for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with chronic, intractable focal pain of the trunk and/or limbs will be screened for participation in this study. Subjects who provide informed consent and meet the eligibility criteria will be enrolled and will undergo a trial procedure. Following the trial phase subjects may receive a permanent implant. Enrollment will continue until 30 subjects receive a permanent implant. We estimate that up to 40 subjects will be enrolled in this registry.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Evoke® therapy neural panel metrics generated by EVA™ | At time of EVA programming and through study completion (up to 30 days)
  The core neural panel metric generated by the Saluda Medical Evoke® therapy system, specifically via its EVA™ sensing technology, is the Evoked Compound Action Potential (ECAP). ECAPs are objective neurophysiological biomarkers that represent the spinal cord's electrical response to stimulation.

SECONDARY OUTCOMES:
Pain Locus of Control | Up to 30 days
  The PLOC classifies the location in which individuals realize predominantly who or what stops the control of their pain. Factor analysis of the main components of this new scale revealed four dimensions: internal LC, chance LC, other people LC (friends and family), doctor and health professional LC. PLOC will be measured using an adapted version of a general purpose, condition-specific Multidimensional Health Locus of Control (MHLC) scale. The responses will be shortened from 6-level to 4-level: strongly agree, agree, disagree and strongly disagree. Each subscale receives an independent score, ranging from 6 to 24 (internal and chance LC subscales) and from 3 to 12 (health professionals and others LC subscales).
Numeric Rating Scale | Up to 30 days
  The NRS is a subjective measure of pain. It is a commonly used pain assessment tool where individuals rate their pain on a scale of 0 to 10, with 0 representing no pain and 10 representing the worst possible pain. It's a simple, quick, and widely accepted method for quantifying pain intensity.
PROMIS-29+2 | Up to 30 days
  The PROMIS-29+2 consists of the PROMIS-29 profile (v2.1) and two PROMIS Cognitive Function Abilities items. The PROMIS-29 is a 29-item profile instrument that assesses 8 universal domains (not disease-specific): Physical Function, Anxiety, Depression, Fatigue, Sleep Disturbance, Ability to Participate in Social Roles and Activities, Pain Interference, and Pain Intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Dustin Reynolds, MD, Principal Investigator — Mount Carmel Health System
Locations (1):
- Mount Carmel Health System, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided